CLINICAL TRIAL: NCT00149903
Title: Multicenter, Double-blind, Randomized, Parallel Group Study on Efficacy and Safety of Enteric-coated Mycophenolate Sodium vs. Mycophenolate Mofetil in de Novo Chinese Renal Transplant Recipients
Brief Title: Study of Enteric-coated Mycophenolate Sodium Versus Mycophenolate Mofetil in Adult de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CERL080A2305
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Mycophenolate sodium (enteric coated)

SUMMARY:
Purpose of study is to compare the efficacy of enteric-coated mycophenolate sodium compared to mycophenolate mofetil in Chinese patients (study conducted in China) as measured by the incidence of biopsy proven acute rejection, graft loss, or death within six months of treatment in de novo renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of first, cadaveric (with donor written consent form) or living related non-HLA identical donor kidney transplant,
* treated with cyclosporine and corticosteroids as primary immunosuppression.

Exclusion Criteria:

* Second or subsequent kidney transplant or multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any other organ
* Patients who have received an investigational drug within four weeks prior to study entry

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-01; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of EC-MPS compared to MMF in Chinese patients as measured by the incidence of biopsy proven acute rejection, graft loss, or death within six months of treatment in de novo renal transplant recipients.

SECONDARY OUTCOMES:
Incidence of biopsy proven acute rejection within six months of treatment in de novo renal transplant recipients
Other variables of efficacy: chronic rejection, graft loss, death.
Safety of EC-MPS as measured by incidence of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- General Hospital, Friendship Hospital, Beijing, No 1 Hospital Peking University, Beijing China; Shanghai No 1 Hospital, Shanghai China; Changzheng Hospital, Shanghai, China; Shanghai Ruij, Beijing, China